CLINICAL TRIAL: NCT02606266
Title: Evaluation of the Benefit of Antiviral Treatment With Valganciclovir on Congenital CMV Infection-related Deafness on Hearing and Balance
Acronym: GANCIMVEAR
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No eligibles patients
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140310; 2015-002232-41 (EudraCT Number)
Record Dates: First submitted 2015-11-05; First posted 2015-11-17 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2018-02

CONDITIONS: Congenital Cytomegalovirus (CMV)
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir; Powders; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valganciclovir (Experimental): Oral valganciclovir (Rovalcyte 50 mg/ml, powder for oral suspension), at a dose of 16 mg/kg 2 times/day (max 900 mg/d) for 6 weeks.
  Interventions: Drug: Valganciclovir
- Control group (No Intervention): Control group with standard care who do not receive the investigational medicinal product

INTERVENTIONS:
Drug: Valganciclovir — Oral valganciclovir (Rovalcyte 50 mg/ml, powder for oral suspension) at a dose of 16 mg/kg 2 times/day (max 900 mg/d) for 6 weeks.
  Other Names: Oral valganciclovir (Rovalcyte 50 mg/ml, powder for oral suspension)
  Arms: Valganciclovir

SUMMARY:
Congenital cytomegalovirus (CMV) infection is the leading cause of non-genetic neurosensory deafness and affects 0.5 to 1% of births. Twenty to thirty per cent of children will develop deafness, some of whom will progress gradually to profound bilateral deafness.

No curative treatment is currently offered for this deterioration in hearing and management involves the use of a hearing aid or cochlear implant. Many studies describe the utility of antiviral treatment on the course of the deafness. These mostly involve neonates with multi-system symptomatic forms of the infection who have been given 6 weeks of ganciclovir possibly switched to valganciclovir, which has shown benefit in stabilising auditory loss, or even improvement.

DETAILED DESCRIPTION:
Congenital cytomegalovirus (CMV) infection is the leading cause of non-genetic neurosensory deafness and affects 0.5 to 1% of births. Twenty to thirty per cent of children will develop deafness, some of whom will progress gradually to profound bilateral deafness.

No curative treatment is currently offered for this deterioration in hearing and management involves the use of a hearing aid or cochlear implant. Many studies describe the utility of antiviral treatment on the course of the deafness. These mostly involve neonates with multi-system symptomatic forms of the infection who have been given 6 weeks of ganciclovir possibly switched to valganciclovir, which has shown benefit in stabilising auditory loss, or even improvement.

ELIGIBILITY:
Inclusion Criteria:

* Children ≥ 6 months old and < 12 years old
* Past history of proven congenital CMV infection
* Auditory threshold of between 40 and 90 dB in at least 1 ear.

Exclusion Criteria:

* Bilateral deafness > 90 dB
* Contraindication to valganciclovir, particularly: Neutropenia with a known neutrophil count of <500/mm3, Hb<8g/dl or platelets< 25,000/mm3 (FBC to be confirmed before randomisation)
* Past history of neutropenia on valganciclovir or allergy to the compound
* Renal impairment with creatinine clearance of < 10 ml/min/1.72m2 (confirmation of renal function before randomisation) according to the Schwartz equation
* Patients on other antiviral treatment
* Gastrointestinal absorption problems
* Patients participating in a biomedical research project on a medicinal product or similar product

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Auditory threshold in db | 6 months

SECONDARY OUTCOMES:
Canal function | 6 months
  Canal function will be assessed using 3 tests : caloric reflex tests; electronystamography & HIT (Head Impulse Test)
FBC (haemoglobin and leukocyte count) | 6 weeks
Serum valganciclovir concentrations | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debré Hospital, Paris, France